CLINICAL TRIAL: NCT05870930
Title: Bioavailability of Phenolic Compounds Following the Consumption of a Carob Beverage
Brief Title: Bioavailability Study of Cretan Carob
Acronym: BIOCRETANCAROB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Responsible Party: Principal Investigator, Andriana C Kaliora, Associate Professor, Harokopio University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CRETAN CAROB_147
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-03

CONDITIONS: Healthy Diet
Keywords: carob; phenolic compound bioavailability; metabolites; bioavailability in humans; Imera carob

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Carob beverage (Experimental)
  Interventions: Other: Carob beverage

INTERVENTIONS:
Other: Carob beverage — Volunteers will consume 2 tablespoons of carob powder in 200mL drinking water.

SUMMARY:
This is an interventional, open-label, single-group, bioavailability postprandial study. The aim of the study is to evaluate the bioavailability of phenolic compounds of a beverage prepared with Cretan carob powder of the Imera cultivar in healthy individuals after consumption.

DETAILED DESCRIPTION:
This is an interventional, open-label, single-group, bioavailability postprandial study. The aim of the study is to evaluate the bioavailability of active constituents of a beverage with carob powder in healthy individuals after consumption. Fifteen apparently healthy male adults of normal body fat mass (non-obese) will be enrolled based on certain inclusion and exclusion criteria. After enrollment, the volunteers will undergo a medical and dietary assessment and will be instructed to follow a low-phytochemical diet (washout) for five consecutive days, excluding from their diet sources of phytochemicals, i.e., fruits, vegetables, legumes, coffee, tea. Compliance with the low-phytochemical diet will be assessed with a 24 h recall during and at the end of the washout period. On the day of the experiment following washout, volunteers will be given a carob beverage (blood samples will be collected 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4-6 h postprandially). Time intervals 0-6h will be used for LC-ESI-MS/MS approach in order to identify putative polyphenol metabolites related to carob consumption.

ELIGIBILITY:
Inclusion Criteria:

* healthy male adults
* normal body fat mass

Exclusion Criteria:

* obesity (according to body fat mass)
* Type 1 Diabetes, cardiovascular diseases, hypertension
* thyroid disorder, liver disease, kidney disease
* gastrointestinal disease
* mental illness
* use of nutraceutical supplements or natural products for weight loss
* dietitians/nutritionists

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-02-10 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Identification of putative polyphenol metabolites related to carob consumption. | Six hours
  Polyphenol metabolites related to carob consumption identified using LC-ESI-MS/MS.

CONTACTS AND LOCATIONS:
Overall Officials: Andriana C Kaliora, Principal Investigator — Harokopio University of Athens, Greece
Locations (1):
- Andriana Kaliora, Athens, Greece

IPD SHARING:
Plan to Share IPD: No